CLINICAL TRIAL: NCT02828761
Title: A Randomized Controlled Trial of Early Coronary Calcium Scoring and Standard Care in Emergency Department Chest Pain Patients
Brief Title: Coronary Calcium Scoring Versus Standard Care for Emergency Department Chest Pain Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never initiated and formally withdrawn with the IRB on 9/14/2023.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-4993
Record Dates: First submitted 2016-06-15; First posted 2016-07-12 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Chest Pain
Keywords: chest pain; calcium score; coronary calcium score; coronary calcium scoring; calcium scoring; cacs; ccs
MeSH Terms: conditions — Chest Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Coronary Calcium Scoring (Experimental): Coronary calcium scoring by multidetector row computed tomography (MDCT).
  Interventions: Device: Coronary Calcium Scoring
- Standard Care (Active Comparator): Standard evaluation of chest pain patient which often includes immediate non-invasive imaging.
  Interventions: Procedure: Standard Care

INTERVENTIONS:
Device: Coronary Calcium Scoring — Scan with 64-detector row or better CT scanners with quantification by the Agatston method.
  Other Names: Calcium Score; Calcium Scoring; Coronary Calcium Score; CACS; CCS
  Arms: Coronary Calcium Scoring
Procedure: Standard Care — Routine clinical monitoring of chest pain patients. Any of a number of non-invasive cardiac tests such as coronary CT angiography, stress echocardiography and stress radionuclide myocardial perfusion imaging may be performed.
  Arms: Standard Care

SUMMARY:
This research asks whether coronary calcium scoring, a non-invasive test based on computed tomography scanning, is a better way to diagnose chest pain patients than other currently used methods. Three of four patients will undergo calcium scoring and the remaining patients will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* complaint of chest pain or pressure
* intermediate risk by HEART score
* clinical indication for non-invasive cardiac imaging
* free of known coronary artery disease

Exclusion Criteria:

* hemodynamic instability
* electrocardiogram suggestive of acute ischemia or myocardial infarction
* unremitting chest pain
* serum troponin levels greater than three times the laboratory threshold
* unable to give his/her own written, informed consent
* pregnant women
* weight > 182 kg
* unable to lie supine for scan
* coronary calcium score, coronary CTA or non-contrast thoracic CT within the last year and available for review
* unable to comply with 30 day follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-09-14 (Estimated); Study Completion 2023-09-14 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 30 days
  number of patients with death, non-fatal heart attack, non-fatal stroke, non-fatal cardiac arrest

SECONDARY OUTCOMES:
Length of Stay | through completion of emergency department stay for each patient, an average of six hours and through completion of hospitalization, an average of two days
  emergency department and inpatient

OTHER OUTCOMES:
Subsequent Major Adverse Cardiovascular Events | minimum of 6 months
  number of patients with death, non-fatal heart attack, non-fatal stroke, non-fatal cardiac arrest
Repeat emergency department visits and hospitalizations | minimum of 6 months
  number of patients with return visits to the emergency department and hospitalizations after the end of the recruitment visit
Subsequent non-invasive cardiac imaging | minimum of 6 months
  number of patients with subsequent stress testing and computed tomography of the heart
Subsequent coronary catheterization | minimum of 6 months
  number of patients with subsequent conventional angiography of the heart
Subsequent percutaneous or surgical coronary revascularization | minimum of 6 months
  number of patients with subsequent coronary angioplasty, coronary stenting and bypass surgery
Total effective radiation dose | minimum of 6 months
  effective radiation dose estimated for procedures involving ionizing radiation
The number of patients reporting changes in aspirin pharmacotherapy | minimum of 6 months
  patients with new prescriptions for or increased dose of aspirin
The number of patients reporting changes in anti-lipid pharmacotherapy | minimum of 6 months
  patients with new prescriptions for or increased dose of lipid lowering medication
The number of patients reporting persistent chest pain on telephone questionnaire | minimum of 6 months
  how many patients report continued chest pain symptoms at follow-up
The number of patients with incidental findings due to imaging and the types of findings | minimum of 6 months
  how many patients had incidental findings on their heart imaging scans

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Levsky, MD, PhD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Montefiore Medical Center - Einstein Division, The Bronx, New York
  - Montefiore Medical Center - Wakefield Division, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No